CLINICAL TRIAL: NCT02093026
Title: An Open-label Study of the Efficacy and Safety of Re-treatments With Rituximab (MabThera®/Rituxan®) in Patients With Active Rheumatoid Arthritis
Brief Title: Extension Study to Assess the Efficacy and Safety of Repeat Treatment With Rituximab (MabThera) in Participants With Active Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WA16855; U2653g (Other: Genentech Inc.)
Record Dates: First submitted 2014-03-19; First posted 2014-03-20 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Methotrexate; Methylprednisolone; Folic Acid

ARMS (1):
- Rituximab (Experimental): Participants will receive rituximab 1 gram intravenously (IV) on Days 1 and 15 of each course of retreatment. In addition, participants will receive methotrexate 10-25 milligrams per week (mg/week) orally or parenterally, methylprednisolone 100 mg IV 30 minutes prior to both rituximab infusions, and a stable dose of folic acid greater than or equal to (>=) 5 mg/week or equivalent. Participants will receive retreatment (next course of rituximab repeat treatment) within 2 weeks of meeting the retreatment criteria as defined in the protocol (minimum of 24 weeks after the first [Day 1] infusion of the last course of rituximab). Repeat treatment will be based on the investigator's decision of prior clinical response to rituximab, clinical need and evidence of active disease (Disease Activity Score in 28 joints >=2.6). Retreatment with rituximab will be continued until withdrawal of consent or study treatment completion on 31 December 2011, whichever is sooner.
  Interventions: Drug: Rituximab; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Folic Acid

INTERVENTIONS:
Drug: Rituximab — Participants will receive rituximab 1 gram IV on Days 1 and 15 of each course of retreatment.
  Other Names: MabThera; Rituxan
Drug: Methotrexate — Participants will receive methotrexate 10-25 mg/week orally or parenterally.
Drug: Methylprednisolone — Participants will receive methylprednisolone 100 mg IV 30 minutes prior to each rituximab infusion.
Drug: Folic Acid — Participants will receive folic acid >= 5 mg/week or equivalent.

SUMMARY:
This study will assess the long-term safety and efficacy of repeat treatment courses of rituximab, in combination with methotrexate in a disease-modifying anti-rheumatic drug (DMARD) inadequate responder population of participants who were previously randomized into studies WA16291 (NCT02693210) or WA17043/U2644g (NCT00074438). The study permits multiple re-treatments until the protocol-defined end-of-treatment date (31 December 2011). Participants will then enter a safety follow-up (SFU) period of at least 48 weeks. This will provide at least 7 years follow-up data on all participants initially randomized into WA16291 or WA17043/U2644g. Approximately 600 participants will potentially be eligible to enter this open label extension study from their respective feeder studies.

ELIGIBILITY:
Inclusion Criteria:

* participants with active RA
* completed 24 weeks of treatment in WA16291 or WA17043
* eligible for re-treatment, based on clinical symptoms (Disease Activity Score in 28 joints >=2.6)
* females of childbearing potential using reliable contraception

Exclusion Criteria:

* participants who participated in rituximab studies WA16291 or WA17043 but withdrew into the safety follow-up phases of these trials
* previous rituximab non-responders
* current treatment with any other disease-modifying drug (apart from methotrexate), or any anti-tumor necrosis factor alfa, anti-interleukin-1, or other biologic therapies
* participants with known active infection of any kind
* evidence of any new or uncontrolled concomitant disease or development of any new contraindications which would preclude repeat treatment with rituximab
* history of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* female participants who are pregnant or breastfeeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2002-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (84):
- United States (39):
  - Birmingham, Alabama
  - Peoria, Arizona
  - Little Rock, Arkansas
  - La Jolla, California
  - Long Beach, California
  - Rancho Mirage, California
  - San Diego, California
  - Colorado Springs, Colorado
  - Aventura, Florida
  - Boca Raton, Florida
  - Fort Lauderdale, Florida
  - Largo, Florida
  - South Miami, Florida
  - Boise, Idaho
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Voorhees Township, New Jersey
  - Great Neck, New York
  - Plainview, New York
  - Rochester, New York
  - Smithtown, New York
  - Greenville, North Carolina
  - Winston-Salem, North Carolina
  - Beachwood, Ohio
  - Dayton, Ohio
  - Mayfield, Ohio
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Duncansville, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Glendale, Wisconsin
  - Wausau, Wisconsin
- Australia (3):
  - Maroochydore, Queensland
  - Melbourne, Victoria
  - Perth, Western Australia
- Ghent, Belgium
- Brazil (3):
  - Curtiba, Paraná
  - Campinas, São Paulo
  - São Paulo, São Paulo
- Canada (4):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - St. John's, Newfoundland and Labrador
  - London, Ontario
- Prague, Czechia
- Finland (2):
  - Heinola
  - Helsinki
- Germany (5):
  - Cologne
  - Leipzig
  - Ratingen
  - Regensburg
  - Würzburg
- Haifa, Israel
- Italy (4):
  - Modena, Emilia-Romagna
  - Udine, Friuli Venezia Giulia
  - Genoa, Liguria
  - Milan, Lombardy
- Mexico (3):
  - Mexico City
  - México
  - Monterrey
- Auckland, New Zealand
- Poland (5):
  - Bialystok
  - Lublin
  - Poznan
  - Warsaw
  - Wroclaw
- Spain (5):
  - Mérida, Badajoz
  - Santiago de Compostela, La Coruña
  - Madrid, Madrid
  - Seville, Sevilla
  - San Cristóbal de La Laguna, Tenerife
- Sweden (2):
  - Gothenburg
  - Stockholm
- United Kingdom (5):
  - Birmingham
  - Cambridge
  - Cannock
  - Leeds
  - Stoke-on-Trent

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included participants who had previously participated in studies WA16291 (NCT02693210) or WA17043 (NCT00074438).
Groups:
- Rituximab: Participants received rituximab 1 gram intravenously (IV) on Days 1 and 15 of each course of retreatment. In addition, participants received methotrexate 10-25 milligrams per week (mg/week) orally or parenterally, methylprednisolone 100 mg IV 30 minutes prior to both rituximab infusions, and a stable dose of folic acid greater than or equal to (>=) 5 mg/week or equivalent. Participants received retreatment (next course of rituximab repeat treatment) within 2 weeks of meeting the retreatment criteria as defined in the protocol (minimum of 24 weeks after the first [Day 1] infusion of the last course of rituximab). Repeat treatment was based on the investigator's decision of prior clinical response to rituximab, clinical need and evidence of active disease (Disease Activity Score in 28 joints >=2.6). Retreatment with rituximab was continued until withdrawal of consent or study treatment completion on 31 December 2011, whichever occurred earlier.
Period: Overall Study
Arm/Group | Rituximab
Started | 465
Completed | 272 (At predefined end-of-treatment date, 272 ongoing participants were designated as completed study.)
Not Completed | 193
Not completed — Adverse Event | 26
Not completed — Death | 10
Not completed — Other | 157

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received any part of an infusion of study medication under Study WA16855.
Groups:
- Rituximab: Participants received rituximab 1 gram IV on Days 1 and 15 of each course of retreatment. In addition, participants received methotrexate 10-25 mg/week orally or parenterally, methylprednisolone 100 mg IV 30 minutes prior to both rituximab infusions, and a stable dose of folic acid >=5 mg/week or equivalent. Participants received retreatment (next course of rituximab repeat treatment) within 2 weeks of meeting the retreatment criteria as defined in the protocol (minimum of 24 weeks after the first [Day 1] infusion of the last course of rituximab). Repeat treatment was based on the investigator's decision of prior clinical response to rituximab, clinical need and evidence of active disease (Disease Activity Score in 28 joints >=2.6). Retreatment with rituximab was continued until withdrawal of consent or study treatment completion on 31 December 2011, whichever occurred earlier.
Arm/Group | Rituximab
Number analyzed (Participants) | 465
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (12.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 364
  Male | 101

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20 (ACR20) Response After First Course
Description: A participant had an ACR20 response if there was at least a 20 percent (%) improvement, ie, reduction from Baseline, in tender joint count (TJC) and swollen joint count (SJC) (28 assessed joints) and in at least 3 of the following 5 parameters: 1) Physician's Global Assessment of Disease Activity [visual analog scale (VAS): 0=no disease activity to 100=maximum disease activity]; 2) Patient's Global Assessment of Disease Activity [VAS: 0=no disease activity to 100=maximum disease activity]; 3) Patient's Assessment of Pain [VAS: 0=no pain to 100=unbearable pain]; 4) Health Assessment Questionnaire [20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do] and 5) an acute-phase reactant (either C-reactive protein [CRP] or erythrocyte sedimentation rate [ESR]). The ACR20 response was compared to Baseline in the precursor studies WA16291 or WA17043.
Time Frame: 24 weeks after first course of rituximab (up to approximately 26 weeks)
Population: Intent to treat (ITT) Population included all participants who received any part of an infusion of study medication under Study WA16855. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 447
percentage of participants | 67.1

2. Primary Outcome: Percentage of Participants With ACR20 Response After Second Course
Description: A participant had an ACR20 response if there was at least a 20% improvement, ie, reduction from Baseline, in TJC and SJC (28 assessed joints) and in at least 3 of the following 5 parameters: 1) Physician's Global Assessment of Disease Activity [VAS: 0=no disease activity to 100=maximum disease activity]; 2) Patient's Global Assessment of Disease Activity [VAS: 0=no disease activity to 100=maximum disease activity]; 3) Patient's Assessment of Pain [VAS: 0=no pain to 100=unbearable pain]; 4) Health Assessment Questionnaire [20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do] and 5) an acute-phase reactant (either CRP or ESR). The ACR20 response was compared to Baseline in the precursor studies WA16291 or WA17043.
Time Frame: 24 weeks after second course of rituximab (median duration of 90.9 weeks)
Population: ITT Population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 384
percentage of participants | 70.8

3. Primary Outcome: Percentage of Participants With ACR20 Response After Third Course
Description: as for outcome 2
Time Frame: 24 weeks after third course of rituximab (median duration of 162.9 weeks)
Population: ITT Population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 310
percentage of participants | 73.2

4. Primary Outcome: Percentage of Participants With ACR20 Response After Fourth Course
Description: as for outcome 2
Time Frame: 24 weeks after fourth course of rituximab (median duration of 232 weeks)
Population: ITT Population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 245
percentage of participants | 75.1

5. Primary Outcome: Percentage of Participants With ACR20 Response After Fifth Course
Description: as for outcome 2
Time Frame: 24 weeks after fifth course of rituximab (median duration of 297.3 weeks)
Population: ITT Population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 175
percentage of participants | 69.7

6. Primary Outcome: Percentage of Participants With ACR20 Response After Sixth Course
Description: as for outcome 2
Time Frame: 24 weeks after sixth course of rituximab (median duration of 354.4 weeks)
Population: ITT Population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 110
percentage of participants | 68.2

7. Primary Outcome: Percentage of Participants With ACR20 Response After Seventh Course
Description: as for outcome 2
Time Frame: 24 weeks after seventh course of rituximab (median duration of 406.7 weeks)
Population: ITT Population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 74
percentage of participants | 59.5

8. Secondary Outcome: Percentage of Participants With ACR50 and ACR70 Response
Description: A participant had an ACR50 and ACR70 response if there was at least a 50% or 70% improvement, ie, reduction from Baseline, in TJC and SJC (28 assessed joints) and in at least 3 of the following 5 parameters: 1) Physician's Global Assessment of disease activity [VAS: 0=no disease activity to 100=maximum disease activity]; 2) Patient's Global Assessment of Disease Activity [VAS: 0=no disease activity to 100=maximum disease activity]; 3) Patient's Assessment of Pain [VAS: 0=no pain to 100=unbearable pain]; 4) Health Assessment Questionnaire [20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do] and 5) an acute-phase reactant (CRP or ESR). The ACR50 and ACR70 responses were compared to Baseline in the precursor studies WA16291 or WA17043.
Time Frame: 24 weeks after first, second, third, fourth, fifth, sixth, and seventh course of rituximab (median duration of 26, 90.9, 162.9, 232, 297.3, 354.4, and 406.7 weeks, respectively)
Population: ITT Population. Here, number of participants analyzed = participants who were evaluable for this outcome. Number analyzed = participants who were evaluable for specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 447
percentage of participants
  ACR50: 24 weeks after first course | 39.4
  ACR50: 24 weeks after second course: number analyzed (Participants) | 384
  ACR50: 24 weeks after second course | 41.9
  ACR50: 24 weeks after third course: number analyzed (Participants) | 310
  ACR50: 24 weeks after third course | 44.8
  ACR50: 24 weeks after fourth course: number analyzed (Participants) | 245
  ACR50: 24 weeks after fourth course | 46.9
  ACR50: 24 weeks after fifth course: number analyzed (Participants) | 175
  ACR50: 24 weeks after fifth course | 40.0
  ACR50: 24 weeks after sixth course: number analyzed (Participants) | 110
  ACR50: 24 weeks after sixth course | 40.0
  ACR50: 24 weeks after seventh course: number analyzed (Participants) | 74
  ACR50: 24 weeks after seventh course | 36.5
  ACR70: 24 weeks after first course | 16.3
  ACR70: 24 weeks after second course: number analyzed (Participants) | 384
  ACR70: 24 weeks after second course | 21.6
  ACR70: 24 weeks after third course: number analyzed (Participants) | 310
  ACR70: 24 weeks after third course | 20.0
  ACR70: 24 weeks after fourth course: number analyzed (Participants) | 245
  ACR70: 24 weeks after fourth course | 20.0
  ACR70: 24 weeks after fifth course: number analyzed (Participants) | 175
  ACR70: 24 weeks after fifth course | 18.9
  ACR70: 24 weeks after sixth course: number analyzed (Participants) | 110
  ACR70: 24 weeks after sixth course | 20.9
  ACR70: 24 weeks after seventh course: number analyzed (Participants) | 74
  ACR70: 24 weeks after seventh course | 18.9

9. Secondary Outcome: American College of Rheumatology Index of Improvement (ACRn) Response
Description: The ACRn is calculated for each participant by taking the lowest percentage improvement in (1) SJC or (2) TJC or (3) the median of the remaining 5 components of the ACR response (patient's assessment of disease activity; patient's global assessment of pain; physician's assessment of disease activity; participant's assessment of physical function; an acute phase reactant value [either CRP or ESR]). The index of improvement in RA, where 0 indicates no improvement and 100 indicates a 100% improvement across all signs and symptoms of RA. ACRn scores were calculated considering the original baseline in the precursor studies WA16291 or WA17043.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 447
units on a scale
  24 weeks after first course | 31.07 (50.188)
  24 weeks after second course: number analyzed (Participants) | 384
  24 weeks after second course | 34.15 (58.769)
  24 weeks after third course: number analyzed (Participants) | 310
  24 weeks after third course | 36.93 (44.912)
  24 weeks after fourth course: number analyzed (Participants) | 245
  24 weeks after fourth course | 39.59 (39.393)
  24 weeks after fifth course: number analyzed (Participants) | 175
  24 weeks after fifth course | 33.76 (48.309)
  24 weeks after sixth course: number analyzed (Participants) | 110
  24 weeks after sixth course | 29.74 (57.197)
  24 weeks after seventh course: number analyzed (Participants) | 74
  24 weeks after seventh course | 24.87 (51.336)

10. Secondary Outcome: Percentage of Participants With Low Disease Activity and Clinical Remission Based on DAS28-ESR
Description: DAS28-ESR was calculated from SJC and TJC using 28 joints count, ESR (millimeters per hour [mm/hour]), and Patient's Global Assessment of Disease Activity (VAS: 0=no disease activity to 100=maximum disease activity). DAS28-ESR = 0.56*square root (sqrt)(TJC28) + 0.28*sqrt(SJC28) + 0.70*natural logarithm (ln) (ESR) + 0.014*Patient's Global Assessment of Disease Activity. Total score range: 0-10, higher score=more disease activity. DAS28-ESR <= 3.2 implied low disease activity (LDA) and DAS28-ESR <2.6 = clinical remission.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 441
percentage of participants
  LDA: 24 weeks after first course | 24.3
  LDA: 24 weeks after second course: number analyzed (Participants) | 382
  LDA: 24 weeks after second course | 30.1
  LDA: 24 weeks after third course: number analyzed (Participants) | 304
  LDA: 24 weeks after third course | 29.3
  LDA: 24 weeks after fourth course: number analyzed (Participants) | 236
  LDA: 24 weeks after fourth course | 28.0
  LDA: 24 weeks after fifth course: number analyzed (Participants) | 172
  LDA: 24 weeks after fifth course | 23.8
  LDA: 24 weeks after sixth course: number analyzed (Participants) | 110
  LDA: 24 weeks after sixth course | 27.3
  LDA: 24 weeks after seventh course: number analyzed (Participants) | 73
  LDA: 24 weeks after seventh course | 24.7
  Remission: 24 weeks after first course | 11.3
  Remission: 24 weeks after second course: number analyzed (Participants) | 382
  Remission: 24 weeks after second course | 16.8
  Remission: 24 weeks after third course: number analyzed (Participants) | 304
  Remission: 24 weeks after third course | 17.1
  Remission: 24 weeks after fourth course: number analyzed (Participants) | 236
  Remission: 24 weeks after fourth course | 15.7
  Remission: 24 weeks after fifth course: number analyzed (Participants) | 172
  Remission: 24 weeks after fifth course | 15.7
  Remission: 24 weeks after sixth course: number analyzed (Participants) | 110
  Remission: 24 weeks after sixth course | 17.3
  Remission: 24 weeks after seventh course: number analyzed (Participants) | 73
  Remission: 24 weeks after seventh course | 13.7

11. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response of 'Good' or 'Moderate'
Description: DAS28-ESR was calculated from SJC and TJC using 28 joints count, ESR (mm/hour), and Physician's Global Assessment of Disease Activity (VAS: 0=no disease activity to 100=maximum disease activity). DAS28-ESR = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.70*ln(ESR) + 0.014*Patient's Global Assessment of Disease Activity. The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders had a change from baseline greater than (>) 1.2 with a DAS28 score less than or equal to (≤) 3.2; moderate responders had a change from baseline >1.2 with a DAS28 score >3.2 to less than or equal to (≤) 5.1 or a change from baseline >0.6 to ≤1.2 with a DAS28 score ≤5.1.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 436
percentage of participants
  Moderate: 24 weeks after first course | 57.8
  Moderate: 24 weeks after second course: number analyzed (Participants) | 378
  Moderate: 24 weeks after second course | 58.5
  Moderate: 24 weeks after third course: number analyzed (Participants) | 299
  Moderate: 24 weeks after third course | 59.5
  Moderate: 24 weeks after fourth course: number analyzed (Participants) | 233
  Moderate: 24 weeks after fourth course | 60.9
  Moderate: 24 weeks after fifth course: number analyzed (Participants) | 169
  Moderate: 24 weeks after fifth course | 62.1
  Moderate: 24 weeks after sixth course: number analyzed (Participants) | 107
  Moderate: 24 weeks after sixth course | 57.0
  Moderate: 24 weeks after seventh course: number analyzed (Participants) | 70
  Moderate: 24 weeks after seventh course | 60.0
  Good: 24 weeks after first course | 24.3
  Good: 24 weeks after second course: number analyzed (Participants) | 378
  Good: 24 weeks after second course | 30.4
  Good: 24 weeks after third course: number analyzed (Participants) | 299
  Good: 24 weeks after third course | 29.1
  Good: 24 weeks after fourth course: number analyzed (Participants) | 233
  Good: 24 weeks after fourth course | 27.9
  Good: 24 weeks after fifth course: number analyzed (Participants) | 169
  Good: 24 weeks after fifth course | 24.3
  Good: 24 weeks after sixth course: number analyzed (Participants) | 107
  Good: 24 weeks after sixth course | 27.1
  Good: 24 weeks after seventh course: number analyzed (Participants) | 70
  Good: 24 weeks after seventh course | 25.7

12. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at 24 Weeks Following Each Course
Description: The HAQ-DI is a questionnaire specific for rheumatoid arthritis and consists of 20 questions referring to 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Participants completed the questionnaire by answering the 20 questions on a scale of 0 (without difficulty) to 3 (unable to do). The total score ranges from 0 (no disability) to 3 (completely disabled). A negative change score indicates improvement.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 447
units on a scale
  24 weeks after first course | -0.51 (0.555)
  24 weeks after second course: number analyzed (Participants) | 386
  24 weeks after second course | -0.48 (0.556)
  24 weeks after third course: number analyzed (Participants) | 309
  24 weeks after third course | -0.43 (0.532)
  24 weeks after fourth course: number analyzed (Participants) | 245
  24 weeks after fourth course | -0.47 (0.529)
  24 weeks after fifth course: number analyzed (Participants) | 174
  24 weeks after fifth course | -0.44 (0.541)
  24 weeks after sixth course: number analyzed (Participants) | 106
  24 weeks after sixth course | -0.38 (0.600)
  24 weeks after seventh course: number analyzed (Participants) | 68
  24 weeks after seventh course | -0.37 (0.576)

13. Secondary Outcome: Change From Baseline in Total Rheumatoid Factors (RF) at 24 Weeks Following Each Course
Time Frame: as for outcome 8
Population: The data for this outcome measure was not analyzed as this outcome was removed per changes in the planned analysis. Per changes in the planned analysis, only key efficacy parameters were analyzed as the long-term efficacy of rituximab is well established.
Arm/Group | Rituximab
Number analyzed (Participants) | 0

14. Secondary Outcome: Percentage of Participants Who Discontinued Treatment Due to Insufficient Response
Time Frame: First, second, third, fourth, fifth, sixth, and seventh course of rituximab (up to a median of approximately 2, 62, 124, 186, 248, 310, and 372 weeks, respectively)
Population: Safety Population. Number analyzed = participants who were evaluable for specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 465
percentage of participants
  First course | 1.1
  Second course: number analyzed (Participants) | 427
  Second course | 2.3
  Third course: number analyzed (Participants) | 350
  Third course | 2.0
  Fourth course: number analyzed (Participants) | 296
  Fourth course | 2.0
  Fifth course: number analyzed (Participants) | 243
  Fifth course | 0.8
  Sixth course: number analyzed (Participants) | 198
  Sixth course | 0.0
  Seventh course: number analyzed (Participants) | 156
  Seventh course | 0.6

15. Secondary Outcome: Time Since Last Treatment Course
Description: Time since last treatment course = The last day of the last dose of rituximab to date of last contact. Date of last contact is the last available date of efficacy, complete medication start date, laboratory, adverse event assessments, early withdrawal visit, date of last contact, or date of death.
Time Frame: Baseline up to 10 years
Population: ITT Population. Here, number of participants analyzed = participants who entered into safety follow-up.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Rituximab
Number analyzed (Participants) | 31
years | 4.21 (2.234)

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 11 years
Description: The rituximab treatment group includes all data beginning with the first treatment with rituximab (either in Study WA17043 or Study WA16291 or Study WA16855). Participants who received placebo are included in the rituximab treatment group from the time they received their first course of rituximab.
Groups:
- Placebo: Data for participants who received placebo in Study WA17043 or WA16291 are included in this reporting group for data collected until they received their first dose of rituximab in this study (Study WA16855). Data from these participants collected after the first dose of rituximab are included in the rituximab reporting group.
Arm/Group | Rituximab | Placebo
Serious Adverse Events (participants affected / at risk) | 230/465 | 12/127
Other Adverse Events (participants affected / at risk) | 422/465 | 93/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=465) | Placebo (N=127)
Pneumonia (Infections and infestations) | 13 | 1
Urinary tract infection (Infections and infestations) | 7 | 0
Lower respiratory tract infection (Infections and infestations) | 6 | 0
Cellulitis (Infections and infestations) | 5 | 0
Bronchopneumonia (Infections and infestations) | 4 | 0
Gastroenteritis (Infections and infestations) | 4 | 0
Respiratory tract infection (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 3 | 0
Urosepsis (Infections and infestations) | 3 | 0
Appendicitis (Infections and infestations) | 2 | 0
Arthritis bacterial (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 2 | 0
Herpes simplex (Infections and infestations) | 2 | 0
Pseudomembranous colitis (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 2 | 0
Pyelonephritis acute (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 2 | 0
Abscess bacterial (Infections and infestations) | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Bursitis infective (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Clostridium difficile sepsis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Epiglottitis (Infections and infestations) | 1 | 0
Gastroenteritis escherichia coli (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Postopeative wound infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection styphlococcal (Infections and infestations) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 19 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 | 0
Joint destruction (Musculoskeletal and connective tissue disorders) | 6 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 2 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degenration (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Still's disease adult onset (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 19 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 4 | 0
Accident (Injury, poisoning and procedural complications) | 3 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 0
Femure fracture (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Myocardial infarction (Cardiac disorders) | 9 | 0
Coronary artery disease (Cardiac disorders) | 5 | 0
Myocardial ischaemia (Cardiac disorders) | 4 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0
Cardiac failure congestive (Cardiac disorders) | 3 | 0
Angina pectoris (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0
Pericarditis (Cardiac disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infaction (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Heart valve incompetence (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Prostrate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Device dislocation (General disorders) | 6 | 0
Chest pain (General disorders) | 4 | 0
Infusion related reaction (General disorders) | 2 | 0
Catheter site haemorrhage (General disorders) | 0 | 1
Death (General disorders) | 1 | 0
Device failure (General disorders) | 1 | 0
Drug interaction (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Umbilical hernia obstructive (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Syncope (Nervous system disorders) | 4 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Cerebral circulatory failure (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cervical myelopathy (Nervous system disorders) | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Serotonin syndrome (Nervous system disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0
Venous thrombosis limb (Vascular disorders) | 2 | 0
Angiopathy (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Rheumatoid vasculitis (Vascular disorders) | 1 | 0
Thromboangiitis obliterans (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 3 | 0
Ovarian cyst (Reproductive system and breast disorders) | 2 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Ovulation pain (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Uterine cervical erosion (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Fatty liver alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 4 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Bladder disorder (Renal and urinary disorders) | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 1 | 0
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Stag horn calculus (Renal and urinary disorders) | 1 | 0
Urethral caruncle (Renal and urinary disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 2 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0
Mesonephric duct cyst (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Basedow's disease (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0
Limb operation (Surgical and medical procedures) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=465) | Placebo (N=127)
Upper respiratory tract infection (Infections and infestations) | 153 | 7
Nasopharyngitis (Infections and infestations) | 145 | 13
Bronchitis (Infections and infestations) | 108 | 6
Urinary tract infection (Infections and infestations) | 102 | 9
Influenza (Infections and infestations) | 56 | 3
Sinusitis (Infections and infestations) | 51 | 1
Pharyngitis (Infections and infestations) | 34 | 5
Gastroenteritis (Infections and infestations) | 31 | 1
Lower respiratory tract infection (Infections and infestations) | 28 | 2
Herpes zoster (Infections and infestations) | 26 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 236 | 54
Back pain (Musculoskeletal and connective tissue disorders) | 84 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 58 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 40 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 32 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 29 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 27 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 | 0
Infusion related reaction (General disorders) | 203 | 25
Oedema peripheral (General disorders) | 45 | 7
Fatigue (General disorders) | 38 | 8
Diarrhoea (Gastrointestinal disorders) | 85 | 9
Nausea (Gastrointestinal disorders) | 62 | 8
Dyspepsia (Gastrointestinal disorders) | 54 | 2
Abdominal pain uppper (Gastrointestinal disorders) | 28 | 2
Abdominal pain (Gastrointestinal disorders) | 26 | 2
Vomiting (Gastrointestinal disorders) | 25 | 3
Headache (Nervous system disorders) | 82 | 9
Dizziness (Nervous system disorders) | 32 | 2
Hypertension (Vascular disorders) | 93 | 6
Depression (Psychiatric disorders) | 41 | 0
Insomnia (Psychiatric disorders) | 29 | 3
Fall (Injury, poisoning and procedural complications) | 64 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 49 | 5
Rash (Skin and subcutaneous tissue disorders) | 43 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 37 | 3
Anaemia (Blood and lymphatic system disorders) | 39 | 0
Cataract (Eye disorders) | 29 | 0
Vertigo (Ear and labyrinth disorders) | 27 | 1

LIMITATIONS AND CAVEATS:
The interpretation of the efficacy data over time should take into consideration that only the response of participants who continued in the study and received further courses of rituximab was captured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.